CLINICAL TRIAL: NCT03618693
Title: The Impact of Perioperative Analgesia in Prostatectomy Patients on Early Quality of Recovery
Brief Title: Impact of Perioperative Analgesia in Prostatectomy Patients on Early Quality of Recovery (SPITALIDO)
Acronym: SPITALIDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUPD01-18
Record Dates: First submitted 2018-07-03; First posted 2018-08-07 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Prostatectomy; Pain
Keywords: prostatectomy; pain; recovery
MeSH Terms: conditions — Pain | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, single centre, interventional, active controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- spinal analgesia SSS (Experimental): Patients will receive a spinal analgesia (group SSS) with a single shot of bupivacaine 0.5% combined with fentanyl intrathecally during induction of anaesthesia. The technique used is referred to daily practice.
  All patients included in the study will receive the same postoperative multimodal analgesia starting at the end of surgery with the following regimen: 30 mg ketorolac 3* per day for 48 hours intravenously and 1 gr 4* per day metamizol intravenously or per oral, depending of the return of bowel function as baseline analgesia during length of hospitalization.
  Additional rescue analgesia will be provided and consisted in boluses of 25 mcg fentanyl intravenously (first 24 hours) and thereafter 5-10 mg oxycodone tablets (per oral administration).
  Postoperative rehabilitation according to the investigators enhanced recovery program including early mobilization and drinking (clear drinks).
  Interventions: Procedure: Spinal anesthesia
- TAP block (Experimental): Patients will receive a TAP block with a single shot of ropivacaine 0.375% combined with clonidine bilaterally. The technique used is referred to daily practice. The blocks will be performed under ultrasound guidance.
  All patients included in the study will receive the same postoperative multimodal analgesia starting at the end of surgery with the following regimen: 30 mg ketorolac 3* per day for 48 hours intravenously and 1 gr 4* per day metamizol intravenously or per oral, depending of the return of bowel function as baseline analgesia during length of hospitalization.
  Additional rescue analgesia will be provided and consisted in boluses of 25 mcg fentanyl intravenously (first 24 hours) and thereafter 5-10 mg oxycodone tablets (per oral administration).
  Postoperative rehabilitation according to the investigators enhanced recovery program including early mobilization and drinking (clear drinks).
  Interventions: Device: TAP Block
- Standard (Active Comparator): Standard care for prostatectomy in the investigators institution consists in the concomitant systemic administration of lidocaine to standard general anaesthesia. Lidocaine will administered initially during induction with a bolus of 1.5 mg per kgBW, followed by an infusion of 1.5 mg per kgBW per hour for 24 hours.
  All patients included in the study will receive the same postoperative multimodal analgesia starting at the end of surgery with the following regimen: 30 mg ketorolac 3* per day for 48 hours and 1 gr 4* per day metamizol intravenously or per oral, depending of the return of bowel function as baseline analgesia during length of hospitalization.
  Additional rescue analgesia will be provided and consisted in boluses of 25 mcg fentanyl intravenously (first 24 hours) and thereafter 5-10 mg oxycodone tablets.
  Postoperative rehabilitation according to the investigators enhanced recovery program including early mobilization and drinking (clear drinks).
  Interventions: Other: Standard

INTERVENTIONS:
Procedure: Spinal anesthesia — Injection of a single shot of local anesthetic bupivacaine 0.5% combined with 20 mcg fentanyl intrathecally.
  Arms: spinal analgesia SSS
Device: TAP Block — TAP block with a single shot of 20ml ropivacaine 0.375% combined with 75 mcg clonidine bilaterally
  Arms: TAP block
Other: Standard — Concomitant systemic administration of lidocaine (as an adjuvant) to the standard general anaesthesia. Lidocaine will administered initially during induction with a bolus of 1.5 mg per kgBW, followed by an infusion of 1.5 mg per kgBW per hour for 24 hours.
  Other Names: Control Intervention
  Arms: Standard

SUMMARY:
The rationale behind this RCT is to assess within 24 hours after surgery the quality of recovery of prostatectomy patients treated with 3 different analgesia concepts (intraoperative spinal analgesia, transversus abdominis plane block, intravenous lidocaine administration) using the quality of recovery (QoR) 15 questionnaire.

DETAILED DESCRIPTION:
Prostatectomy (open or robotic assisted) is a major urological surgery, which is associated with relevant acute postoperative pain. Perioperative analgesic techniques aiming at optimizing postoperative analgesia have to be investigated. Optimal postoperative pain management is one of the key factors leading to enhanced recovery after surgery. Optimal analgesia should aim for optimized patient comfort, fast functional recovery with the fewest side effects thus encouraging the DREAMS concept (DRinking, EAting, Mobilizing and Sleeping).

The perioperative additional use of a spinal single shot analgesia, or a transversus abdominis plane block to general anaesthesia are validated options to enhance pain therapy compared to systemic analgesia alone. However, if the impact on pain scores has been described previously, the impact on the quality of recovery (QoR) is still unclear. Using the assessment of QoR allows for a much more objective and broader assessment of the quality of the postoperative treatment. Indeed, patient's perioperative experience cannot be only focused on pain scores but should involve items like physical independence, patient support, comfort, emotion. All these items are included in already validated QoR questionnaires like the QoR 15 or QoR 40.

The rationale behind this randomized, parallel group, single centre, interventional, active controlled trial is to assess with the QoR 15questionnaire within 24 hours after surgery the quality of recovery of prostatectomy patients treated with 3 different analgesia concepts.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* >18 years old
* eGFR >40ml/min
* Normal liver function
* Prostatectomy (open, robotic assisted)

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Patients with regular use of antiemetics, laxatives, opioids or other types of analgesics
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Severe psychiatric disorder
* Patients with chronic pain
* Preoperative regular use of non-steroidal anti-inflammatory drugs
* Refusal of regional analgesia (SSS or TAP block)
* Contraindication to regional analgesia (SSS or TAP block)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | From preoperative to postoperative day (POD) 1 i.e. within 24 hours after initiation of intervention
  Changes in Quality of Recovery using the validated 15 items quality of recovery (QoR-15) score : QoR is a patient reported outcome short questionnaire that measure the quality of recovery after surgery and anaesthesia. It incorporates 5 dimensions of health (patient support, comfort, emotions, physical independence, pain). This is a shortened validated version of the QoR 40 including 15 items. QoR-15, with a score range from 0 to 150, is easy to perform. Recently a meta-analysis showed that QoR 15 fulfils requirements for outcome measurement instruments.

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting (PONV) | during the first 48 hours postoperatively
  Groups will be assessed for postoperative nausea/vomiting by verbal descriptive scale at 6, 24 and 48 hours respectively.
  Verbal descriptive Scale
  0 No nausea
  1. Mild nausea
  2. Moderate nausea
  3. Frequent vomiting
  4. Severe vomiting
Pain Score | within 6 hours postoperatively, on POD 1 and 2
  Pain will be assessed with the use of pain scores (incisional pain, "deep" visceral pain and pain during coughing/mobilization) according to the validated numeric rating scale (NRS with a range of 0 (no pain) to 10 (maximal pain)).
Gastrointestinal Function | During length of stay, expected to be on average 5 to 7 days
  Return of gastrointestinal function (first flatus, first defecation, tolerance to food) in days.
Opioid Consumption | Within the first 48 hours postoperatively
  Use/amount of opioids intraoperative and postoperatively (transformed in morphine equivalent per 24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wüthrich, MD, Principal Investigator — University Hospital Berne
Locations (1):
- Patrick Wuethrich, Department of Anaesthesiology and Pain Therapy, University Hospital Bern Inselspital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beilstein CM, Huber M, Furrer MA, Loffel LM, Wuethrich PY, Engel D. Impact of analgesic techniques on early quality of recovery after prostatectomy: A 3-arm, randomized trial. Eur J Pain. 2022 Oct;26(9):1990-2002. doi: 10.1002/ejp.2020. Epub 2022 Aug 21. PMID 35960649